CLINICAL TRIAL: NCT03452384
Title: Acupuncture in Depression: From the Clinical Trial, Biomarkers to Molecular Biology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuan-Pin, Chief of psychiatry, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH103-REC2-074
Record Dates: First submitted 2015-05-04; First posted 2018-03-02 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
Keywords: Acupuncture; Traditional chinese medicine; Major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupucture (Experimental): For real acupuncture, disposable acupuncture needles (0.22 x 30-mm sterile stainless needles) were inserted into acupoints for a depth of 10-30 mm in a direction oblique or parallel to the surface.
  Interventions: Other: Acupuncture
- control (Sham Comparator): For sham acupuncture procedure, Streitberger's noninvasive placebo acupuncture needles will be used. Its validity and credibility have been well demonstrated (Streitberger and Kleinhenz, 1998). The needles will be affixed with plastic O-rings and adhesive tapes. The needles with blunt tips will be quickly put onto the same acupoints used in real acupuncture without inserting into the skin.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — For real acupuncture, disposable acupuncture needles (0.22 x 30-mm sterile stainless needles) were inserted into acupoints for a depth of 10-30 mm in a direction oblique or parallel to the surface. To ensure allocation concealment, the inserted needles were affixed with adhesive tapes so that real acupuncture procedure will be identical to control acupuncture procedure. For sham acupuncture procedure, Streitberger's noninvasive placebo acupuncture needles will be used. Its validity and credibility have been well demonstrated (Streitberger and Kleinhenz, 1998).

SUMMARY:
Major depressive disorder (MDD) is a serious psychiatric illness with a high lifetime prevalence rate and causes major clinical, social and economic burden to patients and their family. Despite more than 40 antidepressants with various mechanisms are available on the market, half of patients fail to achieve remission with optimized medication treatment. Due to unsatisfactory efficacy, frequent intolerability and poor compliance of psychopharmacotherapies, novel and safe alternative therapies are critically in need to improve the treatment of depression.

Traditional Chinese medicine (TCM) theory describes a state of health maintained by a balance of energy in the body. If imbalanced, it can be corrected by acupuncture, the insertion of fine needles into different parts of the body. Although there are several clinical trials to demonstrate the antidepressant effects of acupuncture, its biological and physiological mechanisms are still unknown. In addition, clinical depression is frequently accompanied with somatic presentations, which are related to autonomic nervous dysfunction. It would be of interest to know if acupuncture could regulate autonomic nervous system (ANS) and improve the somatic symptoms in depression. The purpose of this study is to assess the effectiveness of acupuncture in the treatment of depression and to determine the influence of acupuncture on the molecular and ANS systems.

DETAILED DESCRIPTION:
In this study,the investigators will test the antidepressant effect of acupuncture versus sham intervention on major depression, in an eight-week, double-blind, randomized-controlled trial in 40 MDD patients who still have significant depressive symptoms without changing at their treatment modality for the last 4 weeks. During the visits at weeks 0 (baseline), 1, 2, 4, 6, 8 (intervention), and 12 (4 weeks after intervention), subjects will be assessed depressive symptoms with the 21-item Hamilton Rating Scale for Depression (HAM-D). Before and after the intervention (Weeks 0 and 8),Computerized TCM constitution diagnosis will be measured and the blood samples will be collected for biomarker analyses, including neurotransmitter, inflammatory molecules and immunologic function. All parts of this research will start after being approved by the Institution Review Board in study sites.

The outcomes of this study could provide the evidence of applying acupuncture as an alternative effective treatment for depression and to improve the understanding of biological mechanisms for its antidepressant effects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of major depressive disorder (MDD)
* Over 18 on the 21-item Hamilton Rating Scale for Depression

Exclusion Criteria:

* Schizophrenia
* Ubstance dependence disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
The Change from Baseline Hamilton depression rating scale at 12 weeks | weeks 0 (baseline) and 12 weeks
  This scale scores 0-64 points;The higher total score indicates a more severe

SECONDARY OUTCOMES:
The Change from Baseline Pittsburgh sleep Quality Inventory rating scale at 12 weeks | weeks 0 (baseline) and 8 weeks
  This scale scores 0-21 points;The higher total score indicates a more severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Kaun-Pin Su, MD, PhD, Principal Investigator — China Medical University Hospital, Tiawan
Locations (1):
- China Medical University Hospital, Taichung, Taiwan